CLINICAL TRIAL: NCT00623038
Title: Trial to Evaluate a Specified Type of APGAR
Acronym: TEST-APGAR
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Prof. Dr. Mario Rüdiger, Dresden University of Technology, Department for Neonatology
Other Study IDs: TEST-APGAR
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Postnatal Condition of a Newborn Infant
Keywords: Apgar score; neonatal assessment; preterm infants; resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is of importance to predict the risk to develop problems after birth. Virginia Apgar developed a score more than 50 years ago that allows a description of the condition of newborns at 1, 5 and 10 minutes after birth. The Apgar score is used for every newborn, however, its applicability is restricted in preterm infants and resuscitated newborns. Thus, two scores have been suggested recently - the Specified Apgar and the Expanded-Apgar score. By combining both scores the Combined-Apgar has been developed as a new delivery room tool.

The purpose of this study is to determine whether the Combined-Apgar predicts poor outcome better than the Specified- or Expanded Apgar alone.

DETAILED DESCRIPTION:
Since the conventional Apgar score has its limitations in preterm or resuscitated infants, specifications of the individual items of the original Apgar score were suggested (Specified Apgar). The Specified-Apgar will slightly change the Apgars' perspective, but will not alter the number of its components. The advantage of the proposed definitions is the applicability in all infants, regardless of resuscitative efforts or gestational age. However, neither the conventional nor the Specified-Apgar score describes the condition of the infant. That problem has been taken up by the American Academy of pediatrics (AAP)and the American College of Obstetricians and Gynecologists (ACOG). They suggested to use an expanded Apgar Score reporting form (Expanded-Apgar)that accounts for concurrent resuscitative interventions. Whereas the Specified-Apgar score describes the condition of the infant, the Expanded-Apgar is a measure of interventions needed to achieve this condition. By combining both scores (Combined-Apgar) the postnatal condition is described in more detail than by a single score alone.

To validate the accuracy of these scores in a population of very preterm infants, the present prospective, observational, international multicenter study is planned. Until today there is no gold standard available to describe infant's conditions and interventions. For the evaluation of the scores it was therefore hypothesized that the Combined Apgar predicts poor outcome (defined as either death or any major morbidity) better than the Specified Apgar or Expanded Apgar alone. Prediction of poor outcome was used as a surrogate parameter to test the predictive value of the Combined-Apgar score in a clinical setting for preterm infants. In an attempt to determine how strong of an association there is between the Combined Apgar Score and neurologic impairment in early childhood, we are presently engaged in a long-term follow-up of all surviving infants at a corrected age of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* gestational age below 32 weeks
* born within the study centres

Exclusion Criteria:

* missing informed consent
* outborn
* major congenital abnormalities
* death in the delivery room

Ages: 1 Minute to 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very preterm infants born prior to 32 completed weeks of gestation
Sampling Method: Probability Sample
Enrollment: 1855 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Poor outcome | Between birth and the day of discharge from first stay in hospital
  Poor outcome is defined as death or the presence of either of the major morbidities: bronchopulmonary dysplasia (BPD), intraventricular hemorrhage (IVH) grade 1-4, cystic periventricular leucomalcia (CPL), retinopathy of prematurity (ROP)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ruediger, Principal Investigator — Department of Neonatology and Pediatric Intensive Care, University Hospital Carl Gustav Carus Dresden, Germany; Helmut Kuester, Principal Investigator — Department of Neonatology and Pediatric Intensiv Care, Ernst-Moritz-Arndt-University Greifswald, Germany

REFERENCES:
- [Derived] Mense L, Nogel S, Kaufmann M, Kuster H, Braun N, Simma B, Rudiger M. Assessing the postnatal condition: the predictive value of single items of the Apgar score. BMC Pediatr. 2025 Mar 19;25(1):214. doi: 10.1186/s12887-025-05565-0. PMID 40102790
- [Derived] Rudiger M, Braun N, Aranda J, Aguar M, Bergert R, Bystricka A, Dimitriou G, El-Atawi K, Ifflaender S, Jung P, Matasova K, Ojinaga V, Petruskeviciene Z, Roll C, Schwindt J, Simma B, Staal N, Valencia G, Vasconcellos MG, Veinla M, Vento M, Weber B, Wendt A, Yigit S, Zotter H, Kuster H; TEST-Apgar Study-Group. Neonatal assessment in the delivery room--Trial to Evaluate a Specified Type of Apgar (TEST-Apgar). BMC Pediatr. 2015 Mar 8;15:18. doi: 10.1186/s12887-015-0334-7. PMID 25884954